CLINICAL TRIAL: NCT05313087
Title: COVID-19 Vaccine Response and Durability In Patients With Chronic Respiratory and Medical Disorders
Brief Title: COVID-19 Vaccine Response in Chronic Respiratory Conditions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Barry Make, Professor of Medicine, National Jewish Health
Other Study IDs: 21-08-054-528
Record Dates: First submitted 2021-06-01; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Controls - who are NOT in any of the groups listed below: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine
- Previous COVID infection: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine
- Asthma receiving immunomodulator medications: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine
- Asthma receiving chronic oral steroids: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine
- Asthma - NOT receiving immunomodulator medications or chronic oral steroids: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine
- Chronic Obstructive Pulmonary Disease (COPD: Adults
  Interventions: Biological: COVID-19 vaccine
- Rheumatoid Arthritis receiving immunomodulator medications: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine
- Rheumatoid Arthritis NOT receiving immunomodulator medications: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine
- Interstitial lung disease: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine
- Cancer patients receiving chemotherapy: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine
- Bronchiectasis: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine
- Cystic fibrosis: Adults and children age 5 and over.
  Interventions: Biological: COVID-19 vaccine

INTERVENTIONS:
Biological: COVID-19 vaccine — assess response to vaccine

SUMMARY:
The investigators will assess the antibody, T cell and B cell responses to SARS-CoV-2 vaccination before and every 3 months for 18 months after the initial vaccination or subsequent vaccinations (boosters) in adults and children including patients with chronic medical conditions.

DETAILED DESCRIPTION:
HYPOTHESES

1. Patients with chronic respiratory diseases will have a lower antibody response to SARS-CoV-2 virus after vaccination and shorter durability of the response than control subjects without chronic disorders.
2. Patients on corticosteroids and other immunomodulator medications for chronic medical disorders will have a lower antibody response to SARS-CoV-2 after vaccination and shorter durability of the response than subjects with chronic disorders who are not being treated with corticosteroids and immunomodulator medications.

SPECIFIC AIMS

1. Enroll up to 1,000 patients receiving a SARS-CoV-2 vaccination (initial or subsequent vaccinations) in an observational study to determine vaccine antibody response and durability.

   1. Obtain blood samples to measure antibody assess the antibody, T cell and B cell responses to SARS-CoV-2 vaccination before and every 3 months for 18 months after the initial vaccination or subsequent vaccinations (boosters) .
   2. Categorize patients by their age, gender, race, ethnicity, underlying chronic disease, disease severity, medical therapy and comorbidities.
   3. Assess the clinical effectiveness of the vaccine to prevent COVID-19 infections.

3. Determine the clinical features and gene expression of patients who are less responsive (have lower antibody levels and shorter duration of antibody response) to SARS-CoV-2 vaccinations.

STUDY DESIGN Patient population - up to 1,000.

Consisting of patients in the following groups:

1. Controls - who are NOT in any of the groups listed below.
2. Previous COVID infection
3. Asthma receiving immunomodulator medications
4. Asthma receiving chronic oral steroids
5. Asthma - NOT receiving immunomodulator medications or chronic oral steroids
6. Chronic Obstructive Pulmonary Disease (COPD)
7. Rheumatoid Arthritis receiving immunomodulator medications
8. Rheumatoid Arthritis NOT receiving immunomodulator medications
9. Interstitial lung disease
10. Cancer patients receiving chemotherapy
11. Bronchiectasis
12. Cystic fibrosis

ELIGIBILITY:
Inclusion Criteria:

* Receipt of a SARS-CoV-2 vaccination

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic medical conditions seen at our medical center (National Jewish Health)
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Antibody response | after SARS-CoV-2 vaccinations
  quantitative spike protein antibody, binding antibody units (BAU)

SECONDARY OUTCOMES:
Antibody change | Change 3 months after vaccinations
  Quantitative spike protein antibody, binding antibody units (BAU)
Antibody change | Change 6 months after vaccinations
  Quantitative spike protein antibody, binding antibody units (BAU)
Antibody change | Change 9 months after vaccinations
  Quantitative spike protein antibody, binding antibody units (BAU)
Antibody change | Change 12 months after vaccinations
  Quantitative spike protein antibody, binding antibody units (BAU)
Antibody change | Change 18 months after vaccinations
  Quantitative spike protein antibody, binding antibody units (BAU)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Make, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be shared once the study results are analyzed and published.
Supporting Information: Study Protocol, CSR
Time Frame: Results will be shared once the study results are analyzed and published.